CLINICAL TRIAL: NCT06452680
Title: The Effect of Preserving Inferior Pulmonary Ligamen on Symptom Burden and Clinical Outcomes in Thoracoscopic Pneumonectomy
Brief Title: The Effect of Preserving Inferior Pulmonary Ligamen on Symptom Burden in Thoracoscopic Pneumonectomy
Acronym: PRO-IPL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, GuiBin Qiao, Professor of Medicine, Guangdong Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KY2023-804-02
Record Dates: First submitted 2024-05-30; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Pulmonary Surgical Procedures; Patient Reported Outcome Measures
Keywords: Inferior pulmonary ligment; Pulmonary Surgical Procedures; Patient Reported Outcome Measures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preservation group (Experimental): In the preservation group, the IPL was untouched
  Interventions: Procedure: Preserving IPL during surgery
- Dissection group (No Intervention): In the dissection group, the IPL was commonly dissected until the inferior pulmonary vein was exposed

INTERVENTIONS:
Procedure: Preserving IPL during surgery — IPL was preserved during surgery
  Arms: Preservation group

SUMMARY:
The investigators conducted a muti-centres randomized controlled clinical trial to explore the effect of preservation of inferior pulmonary ligment compared with dissection.

DETAILED DESCRIPTION:
Dissection of the inferior pulmonary ligament (IPL) has been a common practice in upper lobectomy to facilitate the expansion of the remaining lung, reduce dead space after resection, and minimize complications such as pleural effusion and pulmonary infection. However, studies have found that IPL dissection does not improve patient outcomes. On the contrary, releasing the restriction may lead to excessive movement of the remaining lobes, resulting in significant changes in bronchial angles and lung volume, which can worsen pulmonary function and increase postoperative symptoms. Most existing studies are retrospective, providing relatively low-level evidence. Moreover, previous research has primarily focused on radiographic outcomes and pulmonary function tests results, while the effect on patients' symptom burden has been largely overlooked. From the patient's perspective, symptom burden might be more significant, reflecting the clinical value of changes in radiographic and functional indices. In this study, the investigators applied patient-reported outcomes to measure symptoms. Combined with pulmonary function results and radiological outcomes, the investigators compared the clinical value of preserving versus dissecting the IPL in upper lobectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients underwent upper lobe resection
2. Patients could complete our questionnaires

Exclusion Criteria:

1. Previous history of ipsilateral lung surgery
2. Patients who underwent pleurodesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Cough score postoperation | up to 3 months
  The investigators used PSA-LUNG questionnaire to assess patients symptom burden after surgery. Changing of cough score during 1 month postoperation was chosen as the primary outcome.

SECONDARY OUTCOMES:
Other Symptom burden postoperation PSA-LUNG questionnaire | up to 3 months
  Using PSA-LUNG questionnaire, the investigators assessed shortness of breath, pain, sleeplessness, annoy, and fatigue after surgery.
Radiological outcome | Day 1 after surgery; 1 month after discharge; 3 months after discharge
  Changing of bronchial angels measured with chest x-ray examination or chest CT.
Radiological outcome | Day 1 after surgery; 1 month after discharge; 3 months after discharge
  dead spece rate measured with chest x-ray examination or chest CT.
Radiological outcome | Day 1 after surgery; 1 month after discharge; 3 months after discharge
  degree of lung collapse measured with chest x-ray examination or chest CT.

CONTACTS AND LOCATIONS:
Overall Officials: Guibin Qiao, MD, Study Chair — Guangdong Province People's Hospital
Locations (5):
- China (5):
  - General Hospital of Southern Theater Command of the Chinese People's Liberation Army, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - The Affiliated Panyu Central Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangdong Pharmaceutical University, Guangzhou, Guangdong
  - Shantou University Medical College, Shantou, Guangdong